CLINICAL TRIAL: NCT02632734
Title: Comparison Between CoreBone Coral Particles and CoreBone Coral Cones as Graft After Extraction Sockets for Alveolar Ridge Preservation
Brief Title: The Use of CoreBone Coral Particles vs. Cones for Preservation of Alveolar Bone
Acronym: CoreBone
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Baruch Padeh Medical Center, Poriya (Other Government)
Responsible Party: Principal Investigator, Victoria yaffe gartsbein, Resident in maxillofacial department, The Baruch Padeh Medical Center, Poriya
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CoreBone.CTIL
Record Dates: First submitted 2015-11-08; First posted 2015-12-17 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Bone Loss
Keywords: alveolar bone preservation; coral grafting device
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CoreBone Cone device (Experimental): Experimental: CoreBone Cone device After extraction intervention will include the placement of CoreBone Cone device derived from coral that its dimensions is 4-5mm width and 8-10mm height. One cone for each extraction socket.Its advantage is that it fits well the socket site.Measurements from models taken at different times will be analysed for bone loss. Changes in width and height of alveolar bone will be studied at 3 and 6 month. We predict that CoreBone Cones are more effective than particulate device.
  Interventions: Device: CoreBone Cone device
- CoreBone 500 device (Experimental): After extraction intervention will include the placement of CoreBone500 device derived from coral that is particulate. 0.3-0.5cc for each extraction socket.Its advantage is that it fills well the socket site.Measurements from models taken at different times will be analysed for bone loss. Changes in width and height of alveolar bone will be studied at 3 and 6 month.
  Interventions: Device: CoreBone 500 device

INTERVENTIONS:
Device: CoreBone Cone device — coral derived devices in the form of Cones are placed in extraction sites for preservation of bone during 6month and more.
  Arms: CoreBone Cone device
Device: CoreBone 500 device — coral derived devices in the form of particulate (CoreBone 500) are placed in extraction sites for preservation of bone. Follow up during 6month and more.
  Arms: CoreBone 500 device

SUMMARY:
Normally, dentists do not graft the socket after extraction of teeth. When they do graft they use particulate graft devices. The purpose of this study is to examine whether coral particles of 300-450um in comparison to coral cones of 4-5mm wide and 8-10 mm long will preserve alveolar ridge of maxilla or mandible when grafted immediately after tooth extraction. The coral grafting devices are processed from Porites corals grown in aquariums, under controlled environment. The devices are cleansed and sterilized by gamma irradiation. The measurements during follow ups will be performed from CT x rays and measurements by caliber and models.The width and height measurements from follow up x rays and models. The study will be performed on 10 patients, that two parallel teeth are diagnosed to be extracted, in same patient.The data will be analysed for bone loss and compared to previous published studies. Also comparison between two devices will be performed.

DETAILED DESCRIPTION:
Normally, dentists do not graft the socket after extraction of teeth. When they do graft they use particulate graft devices.The purpose of this study is to examine whether coral particles of 300-450um in comparison to coral cones of 4-5mm wide and 8-10 mm long will preserve alveolar ridge of maxilla or mandible when grafted immediately after tooth extraction.

Methods: 10 patients adults that are diagnosed for extraction of same tooth number ,each on different side of jaw. A non traumatic extraction will be performed, on both sides, sometimes not on same date. After extraction, coral device 'CoreBone500' sterile particles will fill the extraction site. Usually 0.3cc will be used. On the other side of same jaw 'CoreBone' Cone sterile of 4-5mm width and 8-10mm height will be placed in socket. Sutures will be placed and efforts will be put in covering the opening by soft tissues. Follow up of the alveolar ridge preservation will be performed using CT at time of grafting and 6 month later. Measurements during follow ups will be performed by caliber the width and height of alveolar ridge 2 weeks, 3month and 6 month follow up. A clinical follow up of healing soft tissues after grafting and patients complaints of pain will be addressed. If any unusual complaints from patients appears the study will be terminated immediately. From our preclinical studies no adverse effects were found. The analysis of data will be statistically analysed and compared to published data. We expect that CoreBone Cones are more effective in ridge preservation.

ELIGIBILITY:
Inclusion Criteria:

* healthy individuals

Exclusion Criteria:

* smoking
* wound healing is disturbance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Bone loss will be measured from dental impression models of the grafted site by caliper | 2 weeks, 3 month, 6 month after grafting
  The bone loss will be measured from dental impression models of the grafted site that will be taken 2 weeks,3 month,6 month after grafting,using a caliper for measurements from models.

SECONDARY OUTCOMES:
preferred device for socket preservation | 2year
  In addition a comparison between bone loss when CoreBone500 device will be grafted and CoreBone Cone.